CLINICAL TRIAL: NCT07334353
Title: Consensus Guidelines for Pre- and Post-Procedure Skincare in Aesthetic Treatments
Status: Enrolling by invitation | Type: Observational
Sponsor: Venus Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: Pre- and post- procedure care
Record Dates: First submitted 2025-12-09; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Pre and Post Procedure Skin Care; Skin Care
Keywords: Aesthetics; Aesthetic procedures; Skin care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expert Panel: A cohort of dermatology and aesthetic medicine experts participating in a Modified Delphi process to develop consensus recommendations on the pre and post skin care in aesthetic procedures

SUMMARY:
This consensus protocol outlines standardized pre- and post-procedure skincare practices designed to optimize treatment outcomes, enhance skin recovery, and minimize complications following aesthetic procedures. It provides evidence-based guidance for skin preparation before treatment and structured aftercare to support healing, reduce inflammation, prevent infection, and maintain long-term results.

DETAILED DESCRIPTION:
This protocol presents a Delphi-based expert consensus on standardized pre- and post-procedure skincare for aesthetic treatments, developed to optimize clinical outcomes, enhance patient safety, and minimize procedure-related complications. The recommendations apply to a broad spectrum of aesthetic interventions, including injectables, laser and energy-based devices, chemical peels, microneedling, and combination therapies.

Consensus Development Methodology (Delphi Method)

This protocol is developed using the Delphi method, a structured, iterative process designed to achieve expert agreement through multiple rounds of anonymous feedback. A multidisciplinary panel of experienced aesthetic physicians, dermatologists, and skincare experts participates in sequential survey rounds. Each round refines key recommendations based on:

* Aggregated expert responses
* Controlled feedback
* Statistical agreement thresholds

This approach ensures that the final protocol reflects high-level expert agreement, minimizes bias, and supports evidence-informed clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Licensed dermatologists, plastic surgeons, and aesthetic medicine specialists.
* Minimum of five years of clinical experience in aesthetic procedures, including lasers, injectables, chemical peels, or microneedling.
* Demonstrated record of academic or clinical involvement in procedural dermatology or aesthetic medicine.
* Experience managing patients across a range of skin phototypes, particularly Fitzpatrick III-VI.
* Willingness to participate in multiple rounds of survey-based consensus building.
* Commitment to provide independent and anonymous responses

Exclusion Criteria:

* Lack of direct clinical experience with aesthetic procedures.
* Less than five years of relevant clinical practice.
* Inability to commit to all rounds of the Delphi process.
* Conflicts of interest that could bias recommendations (e.g., financial ties to skincare product companies or device manufacturers).
* Insufficient proficiency in the language used for the Delphi survey.
* Failure to complete the initial round, resulting in removal from subsequent rounds.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of an international panel of expert clinicians in aesthetic dermatology and medicine. Participants will include board-certified dermatologists, plastic surgeons, and aesthetic medicine specialists with extensive experience in procedural interventions such as laser therapies, chemical peels, microneedling, and injectable treatments. Eligible experts must have a minimum of five years of clinical practice in aesthetic procedures and a demonstrated record of managing diverse patient populations, including individuals with varying Fitzpatrick skin phototypes (I-VI), with particular attention to skin types III-VI that are more prone to pigmentary complications. Experts will be recruited from academic institutions, professional societies, and clinical practices known for their expertise in aesthetic procedures. The panel is intended to be geographically and ethnically diverse to ensure broad applicability of consensus recommendations. All participants must be
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Level of Expert Consensus on Pre- and Post-Procedure Skincare Protocols for Aesthetic Procedures | 6-8 weeks
  The primary outcomes of this Delphi study are the levels of expert consensus on recommended pre- and post-procedure skincare protocols across various aesthetic procedures. Specifically, the study aims to determine expert agreement on: (1) pre-procedure skin preparation measures, including barrier optimization, hydration, photoprotection, and any topical priming agents; (2) post-procedure care, including barrier repair, management of erythema or inflammation, photoprotection, and timing for reintroduction of active topical agents

CONTACTS AND LOCATIONS:
Locations (1):
- Venus Research Center, Cairo, Egypt